CLINICAL TRIAL: NCT00066547
Title: An Open Label Phase I/II Study of Humanized Human Milk Fat Globule-1 (THEREX) in Patients With Locally Advanced or Metastatic Breast Cancer Following Prior Anthracycline and Taxane Therapy
Brief Title: Monoclonal Antibody Therapy in Treating Women With Locally Advanced or Metastatic Breast Cancer Previously Treated With Combination Chemotherapy
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000316264; UCLA-0212097; ANTISOMA-TOPCAT; ANTISOMA-ASM-THEREX-01
Record Dates: First submitted 2003-08-06; First posted 2003-08-07 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2004-08

CONDITIONS: Breast Cancer
Keywords: recurrent breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — epitumomab

INTERVENTIONS:
Biological: monoclonal antibody HuHMFG1

SUMMARY:
RATIONALE: Monoclonal antibodies can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells.

PURPOSE: Phase I/II trial to study the effect of monoclonal antibody therapy on the body and its effectiveness in treating women who have locally advanced or metastatic breast cancer that was previously treated with combination chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety and tolerability of monoclonal antibody HuHMFG1 in women with locally advanced or metastatic breast cancer previously treated with anthracycline and taxane-based therapy.
* Determine the maximum tolerated dose and appropriate schedule of this drug in these patients.
* Determine the pharmacokinetic profile of this drug in these patients.
* Determine the tumor response rate, progression-free survival, and median survival of patients treated with this drug.
* Analyze immunological markers for evaluation of disease status (e.g., in vitro analysis of antibody-dependent cellular cytotoxicity, natural killer cell activity, complement depletion, and tumor markers CA 15.3 and CEA) in patients treated with this drug.

OUTLINE: This is a dose-escalation, open-label, nonrandomized, multicenter study.

* Phase I: Patients receive monoclonal antibody HuHMFG1 IV over 1-3 hours once every 3 weeks for doses 1 and 2. All subsequent dose intervals are based on individual half-life value of the drug. Patients receive at least 6 doses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of monoclonal antibody HuHMFG1 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

* Phase II:Patients receive monoclonal antibody HuHMFG1 as above at the MTD. Patients are followed at 28 days.

PROJECTED ACCRUAL: Approximately 3-40 patients (3-15 patients for phase I and 19-25 patients for phase II) will be accrued for this study within approximately 12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed breast cancer

  * Locally advanced or metastatic disease
  * No inflammatory breast cancer
* Polymorphic epithelial mucin (PEM) antigen overexpression by immunohistochemistry
* Previously treated with an anthracycline and a taxane in any combination for breast cancer

  * No more than 2 prior chemotherapy regimens, including adjuvant /neoadjuvant therapy
  * No more than 1 prior regimen for distant metastatic disease
  * Any number of prior hormonal or biologic therapy regimens allowed
* Measurable disease

  * At least one unidimensionally measurable lesion not previously irradiated
  * The following are not considered measurable lesions:

    * Bone
    * Leptomeningeal disease
    * Ascites
    * Pleural/pericardial effusion
    * Lymphangitis cutis/pulmonis
    * Abdominal masses not confirmed and followed by imaging techniques
    * Cystic lesions
* No metastases accessible to complete surgical resection
* No CNS metastasis by CT scan
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age

* 18 and over

Sex

* Female

Menopausal status

* Not specified

Performance status

* WHO 0-2

Life expectancy

* At least 4 months

Hematopoietic

* Hemoglobin at least 10 g/dL
* Neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic

* Bilirubin no greater than 1.5 mg/dL
* ALT and AST no greater than 2.5 times upper limit of normal (ULN) (less than 5 times ULN if liver metastases are present)

Renal

* Creatinine no greater than 1.5 times ULN OR
* Creatinine clearance greater than 60 mL/min
* No hyperuricemia (uric acid at least 1.25 times ULN)
* No hypercalcemia (calcium at least 11.5 mg/dL [corrected for serum albumin])

Cardiovascular

* LVEF at least 45% by MUGA or echocardiogram within the past 4 weeks

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3-6 months after study participation
* No other prior malignancy within the past 5 years except adequately treated nonmelanoma skin cancer or cervical intraepithelial neoplasia
* No other concurrent uncontrolled comorbid illness that represents unacceptable risk in the opinion of the investigator
* No legal incapacity

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics
* More than 2 weeks since prior growth factors to aid hematologic recovery
* No other concurrent immunotherapy

Chemotherapy

* See Disease Characteristics
* More than 4 weeks since prior cytotoxic chemotherapy
* No concurrent chemotherapy for metastatic breast cancer

Endocrine therapy

* See Disease Characteristics
* No concurrent endocrine therapy for metastatic breast cancer
* No concurrent chronic corticosteroid therapy
* No concurrent high-dose corticosteroids

Radiotherapy

* More than 4 weeks since prior radiotherapy except for palliation
* No concurrent antitumor radiotherapy except for palliation

Surgery

* More than 4 weeks since prior major surgery

Other

* More than 2 weeks since prior blood transfusions to aid hematologic recovery
* No participation in any other investigational drug study
* No other concurrent investigational drugs
* No other concurrent antitumor therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-05

CONTACTS AND LOCATIONS:
Overall Officials: Mark D. Pegram, MD, Principal Investigator — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California, United States